CLINICAL TRIAL: NCT06924827
Title: A Clinical Study of the Transition of Children From 'Artisanal' Cannabidiol to Epidiolex
Brief Title: A Study to Investigate the Transition of Children From 'Artisanal" Cannabidiol (CBD) to Epidiolex
Acronym: CANN-SWITCH
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Elizabeth Donner (Other)
Collaborators: Jazz Pharmaceuticals (Industry); Alberta Children's Hospital (Other); BC Children's Hospital Research Institute (Other)
Responsible Party: Sponsor-Investigator, Elizabeth Donner, Head, Division of Neurology, The Hospital for Sick Children
Organization: The Hospital for Sick Children (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3524
Record Dates: First submitted 2025-04-04; First posted 2025-04-11 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-03

CONDITIONS: Dravet Syndrome (DS); Lennox-Gastaut Syndrome (LGS)
Keywords: Cannabidiol (CBD); Epidiolex; Seizures; Epilepsy; Lennox-Gastaut Syndrome (LGS); Dravet Syndrome (DS)
MeSH Terms: conditions — Epilepsies, Myoclonic; Lennox Gastaut Syndrome; Seizures; Epilepsy | interventions — Cannabidiol; Solutions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Epidiolex Treatment (Experimental): The participant's dose of Epidiolex will be matched to their dose of 'artisanal' cannabidiol (CBD). Epidiolex will be titrated over two weeks with a concomitant taper of the participant's 'artisanal' CBD. CBD doses during transition week 1 will consist of 75% 'artisanal' and 25% Epidiolex, followed by 50% 'artisanal' and 50% Epidiolex for transition week 2. Participants will commence a CBD dose comprised of 100% Epidiolex once reaching the maintenance period of the study. Participants will remain on their matched dose of Epidiolex throughout the maintenance period, unless a dose modification is clinically indicated for efficacy, safety or tolerability. The daily dose of Epidiolex should not exceed the maximum approved dose of 20 mg/kg/day.
  Interventions: Drug: Epidiolex 100 mg/mL Oral Solution

INTERVENTIONS:
Drug: Epidiolex 100 mg/mL Oral Solution — The participant's 'artisanal' CBD and Epidiolex dose should be taken consistently with food or consistently without food throughout the entire study. The participant's dosing with or without food should be consistent with their method of dosing of 'artisanal' CBD prior to screening. Oral administration is recommended. When necessary, Epidiolex can be enterally administered via silicone feeding tubes, such as nasogastric or gastrostomy tubes.

SUMMARY:
The goal of this clinical trial is to learn the best way to switch children with Lennox-Gastaut Syndrome (LGS) or Dravet Syndrome (DS) taking 'artisanal' (non pharmaceutical-grade) cannabidiol (CBD) to Epidiolex for treatment of seizures. The main questions it aims to answer are:

* How well does a gradual switch from 'artisanal' CBD to Epidiolex work?
* Does the same dose of Epidiolex as 'artisanal' CBD work best?
* What side-effects or medical problems do participants have when switching from 'artisanal' CBD to Epidiolex?

Researchers will examine how successful switching from 'artisanal' CBD to Epidiolex is.

Participants will:

* Gradually increase their dose of Epidiolex and reduce their dose of 'artisanal' CBD until they are taking just Epidiolex
* Visit the clinic five times over 20 weeks for checkups and tests
* Keep a diary of their seizures, symptoms and the number of times they use a rescue seizure medication

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 2 through 18 years, inclusive.
* Clinical diagnosis of Dravet or Lennox Gastaut Syndrome:

Clinical diagnosis of Dravet Syndrome supported by:

1. Onset of seizures within the first year of life.
2. Initial seizures present as fever-induced or fever-triggered seizures, hemi-clonic, generalized tonic-clonic, prolonged seizures (more than 15 minutes).
3. Emergence of other seizure types after 1 year of age.
4. Normal development within the first year of age, then emergence of neurodevelopmental difficulties or delay.

Clinical diagnosis of Lennox Gastaut Syndrome supported by:

a. History of an EEG with slow/disorganized background and slow (<2.5 Hz or less) spike and wave activity or generalized paroxysmal fast activity (GPFA).

b. History of more than 1 type of generalized seizures, including drop seizures (tonic, atonic or tonic-clonic).

* Participant must be willing and able to give written informed consent for participation. If the participant is not qualified or unable to provide written consent based on age, development, intellectual capacity or other factors, the parent or legally authorized representative must provide written informed consent on their behalf.
* Must be on a stable dose of a licensed artisanal cannabidiol (CBD) product as maintenance therapy for seizure control for a minimum of 3 months prior to screening (visit 1).
* 'Artisanal' CBD dose must be between 5 mg/kg/day and 20mg/kg/day.
* 'Artisanal' CBD preparation must be a high CBD to THC formulation defined as a minimum CBD:THC ratio of 20:1.
* Must be taking a minimum of 1 other anti-seizure medication (ASM) in addition to an 'artisanal' form of CBD.
* Must be on a stable dose of ASMs for a minimum of 28 days prior to screening (visit 1) and remain on a stable dose throughout the entire study unless medically necessary change(s) are required for safety events.
* Participants with a vagal nerve stimulator (VNS) must have the following conditions met:

  1. The VNS has been in place for a minimum of 3 months prior to screening (visit 1).
  2. The settings have remained constant for 28 days prior to screening (visit 1) and are expected to remain constant throughout the entire study.
  3. The battery is expected to last for the duration of the study.
* Participants on the ketogenic diet must be on a stable regime for a minimum of 28 days prior to screening (visit 1) and expected to remain stable throughout the entire study.
* Participant and/or caregiver must be willing to maintain a seizure diary throughout the duration of the study.

Exclusion Criteria:

* Previous or current exposure to Epidiolex.
* Supplemental use of cannabinoid-containing products, including but not limited to:

  1. Recreational use of cannabis.
  2. Use of artisanal CBD as a seizure rescue medication.
  3. Use of more than one formulation of 'artisanal' CBD (e.g. THC supplementation).
* Pregnant or breastfeeding.
* Any clinically significant, unstable medical condition other than epilepsy that, in the opinion of the investigator, could place the participant at increased risk or interfere with the results of the study.
* Hepatic impairment at screening (visit 1) defined as either of the following conditions:

  1. ALT or AST > 5x upper limit of normal (ULN).
  2. ALT or AST > 3x ULN and total bilirubin >2x ULN (or international normalized ratio >1.5).
* Known sensitivity to any ingredient in Epidiolex, including sesame and sesame oil.
* Unwillingness to refrain from alcohol consumption throughout the duration of the study.
* Unwillingness of females of childbearing potential to use a highly effective form of birth control. Acceptable methods include: hormonal contraceptives, intra-uterine devices, bilateral tube occlusion, vasectomized partner and sexual abstinence.
* Currently enrolled in another clinical trial.
* Have suicidal plan/intent, active suicidal thoughts, or a suicide attempt in the past 6 month prior to screening.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 25 (Estimated)
Dates: Start 2026-02-02 (Estimated); Primary Completion 2028-02-02 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
The success rate of transition of children from 'artisanal' CBD to Epidiolex. | Baseline (visit 2, Day 1) through visit 4 (Day 15), the two-week transition phase.
  Participants successfully transitioned from 'artisanal' CBD to Epidiolex if they complete the transition protocol and continue treatment with Epidiolex at visit 2 following the two-week transition phase of the study. The success rate will be determined as the percentage of participants that complete the two-week transition phase.

SECONDARY OUTCOMES:
The acceptability rate of Epidiolex in children previously treated with 'artisanal' CBD. | Baseline (visit 2, Day 15) to end of treatment (visit 7, Day 85).
  Participants accepted transition to Epidiolex if they continued treatment with Epidiolex after the last scheduled visit of the maintenance period (visit 7). The acceptability rate will be determined as the percentage of participants that continue treatment with Epidiolex after the last scheduled visit of the maintenance period (visit 7, Day 85).
The change in seizure frequency following transition of children from 'artisanal' CBD to Epidiolex. | Baseline (visit 2, Day 1) through the end of treatment (visit 7, Day 85).
  The percent change (increase or decrease) from baseline in 28-day seizure frequency during the maintenance period. Seizure frequency will be calculated as the total number of seizures divided by the number of days with seizure data, multiplied by 28.
Change in reported Pediatric Epilepsy Side-Effects Questionnaire (PESQ) score. | Baseline (visit 2, Day 1) through visit 4 (Day 15), visit 5 (Day 29) and end of treatment (visit 7, Day 85).
  The Pediatric Epilepsy Side Effects Questionnaire (PESQ) is a rating scale to assess pediatric participant-reported side effects associated with anti-seizure medication treatment. Each side-effect is rated on a 6-point Likert scale as follows: (1) - "Not present", (2) - "Low severity", (3) - "Low-moderate severity", (4) - "Moderate severity", (5) - "Moderate-high severity", (6) - "High severity". Higher scores indicated worse side-effects.
Change Clinical Global Impression of Improvement (CGI-I) score. | Baseline (visit 2, Day 1) through visit 5 (Day 29) and end of treatment (visit 7, Day 85).
  The Clinical Global Impression of Improvement (CGI-I) is a 7-point Likert scale used to rate the overall change in seizure control, behaviour, safety and tolerability after transitioning to Epidiolex relative to baseline. The participant's overall improvement is rated by the clinician and caregiver as: 1- "very much improved", 2- "much improved', 3- "minimally improved", 4- "no change", 5- "minimally worse", 6- "much worse", and 7- "very much worse". Higher scores indicate worse condition.
Change in Clinical Global Impression of Seizure Intensity/Duration (CGI-CSID) score. | Baseline (visit 2, Day 1) through visit 5 (Day 29) and end of treatment (visit 7, Day 85).
  The Clinical Global Impression of Change in Seizure Intensity/Duration (CGI-CSID) is a 7-point Likert scale used to rate the overall change in seizure intensity and/or duration after transitioning to Epidiolex relative to baseline. The participant's overall improvement is rated by the clinician and caregiver as: 1- "very much improved", 2- "much improved', 3- "minimally improved", 4- "no change", 5- "minimally worse", 6- "much worse", and 7- "very much worse". Higher scores indicate worse condition.
Change in Quality of Life in Childhood Epilepsy Questionnaire (QOLCE-55) score. | Baseline (visit 2, Day 1) through end of treatment (visit 7, Day 85).
  The Quality of Life in Childhood Epilepsy Questionnaire (QOLCE-55) is a caregiver-reported questionnaire that evaluates quality of life in epileptic children. It contains 55 questions that measure quality of life in 4 areas: cognitive functioning, emotional functioning, social functioning, and physical functioning. Each question is rated on a 5-point Likert scale, with the option to answer "not applicable" as follows: (1) - "All of the time", (2) - "Most of the time", (3) - "Some of the time", (4) - "A little of the time", (5) - "None of the time", (6) - Not applicable. Higher scores indicate higher health-related quality of life.
Change in Measure Yourself Medical Outcome Profile 2 (MYMOP2) score. | Baseline (visit 2, Day 1) through end of treatment (visit 7, Day 85)
  The Measure Yourself Medical Outcome Profile 2 (MYMOP2) questionnaire is a scale that allows participants or caregivers to identify the problem(s) that are most important to them/the participant, and rate the severity of the problem (s) on a 7-point Likert scale ranging from 0 (as good as it can be) to 6 (as bad as it could be). Higher scores indicate worse problems.
Change in Children's Sleep Habit Questionnaire (CSHQ) score. | Baseline (visit 2, Day 1) through visit 5 (Day 29) and end of treatment (visit 7, Day 85).
  The Children's Sleep Habit Questionnaire (CSHQ) is a caregiver-reported questionnaire to measure sleep behaviours in children. The questionnaire has 45 questions about bedtime resistance, sleep onset delay, sleep duration, sleep anxiety, night wakings, parasomnias, sleep disordered breathing, and daytime sleepiness. Each question is rated on a 3-point Likert scale as follows: (1) - "Usually (5 or more times in a week)", (2) - "Sometimes (2-4 times in a week)", (3) - Rarely (never or 1 time during a week). A higher score indicates more sleep problems.
Number of dose increases in anti-seizure medications (ASMs) after starting Epidiolex. | Baseline (visit 2, Day 1) through end of treatment (visit 7, Day 85).
  The number of dose increases in anti-seizure medications (ASMs), including Epidiolex, due to worsening seizure burden or other factors.
Number of dose decreases in anti-seizure medications (ASMs) after starting Epidiolex. | Baseline (visit 2, Day 1) through end of treatment (visit 7, Day 85).
  The number of dose increases in anti-seizure medications (ASMs), including Epidiolex, due to adverse events or other factors.
Frequency of adverse events of special interest (AESIs) after starting Epidiolex. | Baseline (visit 2, Day 1) through end of treatment (visit 7, Day 85).
  Adverse events of special interest (AESIs) include: somnolence, sedation, appetite changes, gastro-intestinal upset (including diarrhea and vomiting), and transaminase elevations. Frequency of AESIs will be measured by determining the total number of AESIs experienced throughout the treatment period of the study.
Severity of adverse events of special interest (AESIs) after starting Epidiolex. | Baseline (visit 2, Day 1) through end of treatment (visit 7, Day 85).
  Adverse events of special interest (AESIs) include: somnolence, sedation, appetite changes, gastro-intestinal upset (including diarrhea and vomiting), and transaminase elevations. The severity of AESIs will be assessed as: "Mild - Events require minimal or no treatment and do not interfere with the participant's daily activities", "Moderate - Events result in a low level of inconvenience or concern", or "Severe - Events interrupt a participant's usual daily activity and may require therapy or other treatment". The total number of mild, moderate and severe AESIs experienced throughout the treatment period of the study will be determined.
Duration of adverse events of special interest (AESIs) after starting Epidiolex. | Baseline (visit 2, Day 1) through end of treatment (visit 7, Day 85).
  Adverse events of special interest (AESIs) include: somnolence, sedation, appetite changes, gastro-intestinal upset (including diarrhea and vomiting), and transaminase elevations. The duration of AESIs will be measured by calculating the length of individual AESIs experienced throughout the treatment period of the study.
Withdrawal rate due to adverse events after starting Epidiolex. | Baseline (visit 2, Day 1) through end of treatment (visit 7, Day 85).
  The withdrawal rate will be determined as the percentage of participants who withdraw from the study and discontinue Epidiolex due to adverse events.
The change in frequency of seizure rescue medication use following transition from 'artisanal' CBD to Epidiolex. | Baseline (visit 2, Day 1) through end of treatment (visit 7, Day 85).
  The percent change (increase or decrease) from baseline in 28-day seizure rescue medication use during the maintenance period. Rescue medication frequency will be calculated as the total number of doses of rescue medication administered divided by the number of days with diary data, multiplied by 28.
Change in Columbia-Suicide Severity Rating Scale (C-SSRS) score. | Baseline (visit 1, Day -28) through end of treatment (visit 7, Day 85).
  The Columbia-Suicide Severity Rating Scale (C-SSRS) assess the risk of suicidal ideation and behaviour. The questions are divided into categories related to ideation (thoughts) and behaviour (actions). Higher scores indicate more serious/worse suicidal ideation or behaviors.

OTHER OUTCOMES:
Change in Short Form 12 (SF-12) score. | Baseline (visit 2, Day 1) through end of treatment (visit 7, Day 85).
  The Short Form 12 (SF-12) is a survey designed to assess health and well-being from a self-perspective. The questionnaire is a 12-item measure evaluating 8 areas of health: physical functioning, physical and emotional limitations, social functioning, bodily pain, general and mental health. The questionnaire will be administered to the caregiver. Higher scores represent better health-related quality-of-life.
Motivation for switching from 'artisanal' CBD to Epidiolex. | Baseline (visit 1, Day -28), once at beginning of study.
  The switching questionnaire consists of two multiple choice questions, along with an open-ended question designed to understand the caregiver's primary and secondary reasons for transitioning their child from 'artisanal' CBD to Epidiolex.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Donner, MD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada